CLINICAL TRIAL: NCT04014504
Title: Effect of Pethidine Analgesia on False Positivity in Neonatal Hearing Screening Test
Brief Title: Pethidine Analgesia and Neonatal Hearing Screening Test
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.07.07
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Hearing Loss; Newborn Complication
Keywords: Newborn Hearing Screening; Otoacoustic emissions; Pethidine; False positive
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The results of the hearing screening test of the beats of the patients who have undergone pethidine in the active phase of labor will be examined. the results will be reported as passed - remained; the false positivity rate according to the retest of the remaining group is to be looked at.
  Interventions: Diagnostic Test: Neonatal Hearing Screening Test
- control group: In the active phase of labor, hearing screening test results of beats of pediatric patients will be evaluated. the results will be reported as passed - remained; the false positivity rate according to the retest of the remaining group is to be looked at. control group.
  Interventions: Diagnostic Test: Neonatal Hearing Screening Test

INTERVENTIONS:
Diagnostic Test: Neonatal Hearing Screening Test — neonatal hearing screening test results will be evaluated.

SUMMARY:
Neonatal hearing screening may fail due to some perinatal and neonatal factors. It is well known that false positivity in newborn hearing screening increases cost and maternal anxiety and anxiety. There is still widespread concern about the use of opoid analgesics to relieve pain during labor. The aim of this study was to determine the effects of pethidine administered during labor on neonatal hearing screening test false positivity rates.

DETAILED DESCRIPTION:
The study group consisted of patients receiving 50 mg intramuscular (I.M) pethidine at the beginning of the active phase of labor and the control group consisted of patients not receiving pethidine. Newborns were evaluated by otoacoustic emission (OAE) test. The OAE test was performed before the patients were discharged. Perinatal and neonatal variables and test results were recorded and the relationship between false positivity and pethidine use was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* term singleton pregnancy,
* Gave birth at 37-41 weeks of gestation,
* without chronic internal disease,
* Pregnant women were included in the study.

Exclusion Criteria:

* Newborn hospitalized in intensive care,
* congenital / chromosomal anomaly,
* congenital CMV infection,
* facial / ear deformities,
* family with hearing problems,
* those with hyperbilirunemia,
* tested at <12 hours after birth,
* maternal infection,
* Diabetes mellitus, recurrent abortion,
* smoking,
* plesanta previa,
* prolonged premature rupture of the membrane (more than 12 hours), epidural -analgesia and
* newborns who were at risk of asphyxia hypoxia were excluded from the study.

Ages: 24 Hours to 14 Days | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: term singleton pregnancy,Gave birth at 37-41 weeks of gestation, without chronic internal disease,Pregnant women were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Hearing Screening Test | 2 week
  neonatal hearing screening test results will be evaluated. will be reported as left or passed.
  The "pass'' en response observed in the hearing screening device indicates that the baby passed the screening test, and the" refer "response indicates that the baby has failed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)